CLINICAL TRIAL: NCT01137721
Title: State Of The Art Functional Imaging In Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SCDMR4
Record Dates: First submitted 2010-06-03; First posted 2010-06-04 (Estimated); Last update posted 2018-08-23 (Actual); Status verified 2016-08

CONDITIONS: Sickle Cell Anemia
Keywords: magnetic resonance imaging; sickle cell disease; hydroxyurea therapy
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Pre-Hydroxyurea - subjects with SCD: Patients with a diagnosis of HbSS (sickle cell anemia) or HbS/ß0-thalassemia (beta thalassemia) who will be treated with hydroxyurea therapy.
- Sibling control: Sibling control with no diagnosis of HbSS or HbS/ß0-thalassemia.
- Observational - subjects with SCD: Patients with a diagnosis of HbSS or HbS/ß0-thalassemia.
- Pre-transfusion - subjects with SCD: Patients with a diagnosis of HbSS or HbS/ß0-thalassemia who will be treated with transfusion therapy.

SUMMARY:
Sickle cell anemia (SCA) is a serious blood disease with blood vessel changes leading to brain injury and stroke. Studies show about 11% of patients with SCA will develop obvious stroke before age 20 years, with children less than 10 years of age especially vulnerable. The main objective of the SCDMR4[State Of The Art Functional Imaging In Sickle Cell Disease] trial is to compare the gray matter cerebral blood flow, measured by MRI,[magnetic resonance imaging] ASL [Arterial Spin Labeling] perfusion before treatment begins and after the appropriate hydroxyurea dosage is reached (~ one year). Other important objectives of the SCDMR4 trial include describing the effect of hydroxyurea therapy and transfusion therapy on the functional MRI response, diffusion tensor imaging of white matter, brain function, and transcranial Doppler blood velocities.

DETAILED DESCRIPTION:
The Primary Objective of the study is to compare the research participant's GM [Gray Matter] CBF [Cerebral Blood Flow] by ASL [Arterial Spin Labeling] techniques before and after reaching a stable hydroxyurea MTD [Maximum Tolerated Dose] (12±3 months after starting hydroxyurea).

This is an observational study. Participants receive hydroxyurea as part of their standard of care treatment. This study will observe the above measures prior to beginning hydroxyurea and after participants reach the maximum tolerated dose in order to describe the effect of therapy on the participants' functional response.

ELIGIBILITY:
Inclusion Criteria for Pre-Hydroxyurea or Pre-Transfusion Therapy Study Participants:

1. The diagnosis of HbSS or HbS/ß0-thalassemia
2. Age: 8.0 -- <19 years old

Inclusion Criteria for Study Participants for Observation:

1. The diagnosis of HbSS or HbS/ß0-thalassemia
2. Age: 8.0 -- <19 years old

Inclusion Criteria for Study Participants for Family Related Controls:

1. No diagnosis of HbSS or HbS/ß0-thalassemia
2. Age: 8.0 -- <19 years old

Exclusion Criteria for Pre-Hydroxyurea or Pre-Transfusion Therapy Study Participants:

1. Unable to tolerate the anatomical or fMRI [functional magnetic resonance imaging] without sedation or anesthesia
2. Currently receiving hydroxyurea therapy or transfusion therapy
3. Previous stem cell transplant or other myelosuppressive therapy
4. History of clinical stroke
5. Inability or unwillingness of research participant or legal guardian/representative to give written informed consent/assent.

Exclusion Criteria for Study Participants for Observation:

1. Unable to tolerate anatomical or fMRI components without sedation or anesthesia
2. Currently receiving hydroxyurea or transfusion therapy
3. Previous stem cell transplant or other myelosuppressive therapy
4. History of clinical stroke
5. Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Exclusion Criteria for Study Participants for Family Related Controls:

1. Unable to tolerate anatomical or fMRI components without sedation or anesthesia
2. Currently receiving hydroxyurea or transfusion therapy
3. Previous stem cell transplant or other myelosuppressive therapy
4. History of clinical stroke
5. Inability or unwillingness of research participant or legal guardian/representative to give written informed consent.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The potential research participants will be recruited, screened and consented from the School-Age and Teen Sickle Cell Clinics by the referring St. Jude hematology co-investigators. There will be no advertisement per se. Affiliate hematology co-investigators will contact St. Jude hematology co-investigators about potentially eligible research participants. Affiliate potential research participants will be screened, and if appropriate, consented and tested at St. Jude institution.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2010-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Change in cerebral blood flow | from baseline to 12 +/- 3 months
  Change in gray matter cerebral blood flow measured by arterial spin labeling techniques from before (baseline) to after reaching a stable hydroxyurea maximum tolerated dose.

SECONDARY OUTCOMES:
Change in cerebral blood flow by territory | From baseline to 12 +/- 3 months
  Change in gray matter cerebral blood flow in individual anterior cerebral artery, middle cerebral artery, and posterior cerebral artery territories, and hemispheric gray matter measured by arterial spin labeling techniques from before (baseline) to after reaching a stable hydroxyurea maximum tolerated dose.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Ogg, M.D, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols